CLINICAL TRIAL: NCT04138511
Title: Ecofisio, a Mobile Application for Assessment and Diagnosis Using Ultrasound Imaging for Undergraduate Health Science Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irene Cantarero Villanueva (Other)
Responsible Party: Sponsor-Investigator, Irene Cantarero Villanueva, Principal Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EcoFisio PID 14-56
Record Dates: First submitted 2019-10-18; First posted 2019-10-24 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Sport Injury; Educational Problems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (ECOFISIO) (Experimental): Ecofisio Group received the ECOFISIO mobile application after students had received theoretical-practical lessons about ultrasound skills in sports pathologies areas, to study the subject.
  Interventions: Device: ECOFISIO
- Control Group (No Intervention): Students received theoretical-practical lessons about ultrasound skills in sports pathologies areas and used traditional study models, to study the subject

INTERVENTIONS:
Device: ECOFISIO — The ECOFISIO application is focused on sports pathologies and contains relevant written and digital information about ultrasound imaging and managing as well as diagnosis of sport injuries.
  Arms: Experimental group (ECOFISIO)

SUMMARY:
The new called "Generation Z" is starting to reach college age. They have adopted technology and create a deep dependence on it, becoming more drawn to the virtual world. M-learning has experienced a huge expansion in recent years in both, medical context and medical and health's sciences education. Ultrasound is an important diagnosis technique in physiotherapy, especially in sports pathology. m-Learning environments could be a useful tool for improve the comprehension of ultrasound concepts and the acquisition of professional competencies. The purpose of this study was to evaluate the efficacy and the use of an interactive platform accessible through mobile devices (ECOFISIO) using ultrasound imaging for the development of professional competencies in the evaluation and diagnosis of sports pathologies.

Participants were 110 undergraduate students enrolled in two groups of this randomized controlled multicentre study: a control group (traditional learning) and experimental group (ECOFISIO mobile application). All participants were assessed both theoretically and by means of the Objective Structured Clinical Examination (OSCE) exams.

ELIGIBILITY:
Inclusion criteria:

* To have anatomy and biomechanics previous knowledge.
* To be enrolled in any required subject.
* To have basic ability to use a mobile application.
* To have a smartphone with Internet Access (Android Operating System).

Exclusion criteria:

- To have received any previous training in ultrasound imaging and managing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Objective Structured Clinical Examination (OSCE) | After the self-study periods in both study groups, up to two weeks.
  An OSCE is a type of examination often used in health sciences. It is designed to test clinical skill performance and competence in a range of skills. The OSCE content and scoring procedures are standardized. It consists of five stations with five specific components of musculoskeletal ultrasound. Each test station is designed to focus on an area of clinical competence, namely: patient positioning, ultrasound probe positioning, ultrasound probe orientation (angle), ultrasound probe management and image adjustment. A standardized scoring tool is used to record what you do or don't do well, with a Likert scale with a range of 0 to 4 to rate the specific efficiency of each component. All OSCE candidates experience the same problem and are asked to perform the same task, within the same deadline. OSCEs are now widely used in undergraduate, graduate and undergraduate assessments. Overall reliability for this tool, Cronbach's alpha, is 0.89.

SECONDARY OUTCOMES:
Multiple Choice Questionnaire (MCQ) | After the self-study periods in both study groups, up to two weeks.
  The MCQ is an evaluation of the theoretical knowledge with 20 questions where a maximum score of 10 points could be obtained.The higher score, the better outcome.

OTHER OUTCOMES:
Satisfaction survey | After the self-study periods in both study groups, up to two weeks.
  a specific 5-point Likert questionnaire (from 1 indicating 'disagree' to 5 indicating 'strongly agree'), which had been used in similar contexts previously

REFERENCES:
- [Derived] Lozano-Lozano M, Galiano-Castillo N, Fernandez-Lao C, Postigo-Martin P, Alvarez-Salvago F, Arroyo-Morales M, Cantarero-Villanueva I. The Ecofisio Mobile App for Assessment and Diagnosis Using Ultrasound Imaging for Undergraduate Health Science Students: Multicenter Randomized Controlled Trial. J Med Internet Res. 2020 Mar 10;22(3):e16258. doi: 10.2196/16258. PMID 32154784